CLINICAL TRIAL: NCT00745043
Title: Do Beta-blockers Affect the Use of Beta-agonist Inhalers in COPD?
Brief Title: Beta-Blocker in Chronic Obstructive Pulmonary Disease (COPD) Study
Acronym: BOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Waikato Hospital (Other)
Collaborators: Waikato Hospital Research Fund (Unknown)
Responsible Party: Dr Catherina Chang Research Fellow, Respiratory Research Waikato Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NTX/05/04/035
Record Dates: First submitted 2008-08-29; First posted 2008-09-01 (Estimated); Last update posted 2024-07-29 (Actual); Status verified 2008-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Betablockers; bronchodilator; exercise capacity; methacholine challenge
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- R302 (Placebo Comparator): Daily placebo capsules
  Interventions: Drug: bronchodilator response
- R303 (Active Comparator): Daily metoprolol 95mg capsules
  Interventions: Drug: bronchodilator response
- R304 (Active Comparator): Daily propranolol 80mg capsules
  Interventions: Drug: bronchodilator response
- Open Label (Active Comparator): Daily Metoprolol 190mg capsules
  Interventions: Drug: bronchodilator response

INTERVENTIONS:
Drug: bronchodilator response

SUMMARY:
Smoking causes both smoking related lung disease (COPD) and ischaemic heart disease. These are very common conditions and many patients have both diseases. Beta-blocker drugs are extensively used in the treatment of angina, high blood pressure and after heart attacks to decrease symptoms and prolong life. Beta-agonists are used in COPD to decrease breathlessness and improve exercise tolerance. It used to be thought that beta-blockers cannot be used in COPD patients as they may make the breathlessness worse, but it has now been established that they can be used safely. Beta-blocker drugs and beta-agonists have 'opposite' effects on the body and the investigators do not know if they can work together or if they would cancel each other out. The investigators also do not know which of the different types of beta-blockers now available are better for COPD patients. This study will investigate what happens to the airways of people taking both of these drugs.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* > 40 years of age
* > 15 pack year smoking history

Exclusion Criteria:

* Contra-indication to beta-blocker use
* Severe COPD FEV1 < 30% or 1 L
* Not responsive the methacholine

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-05; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Bronchodilator response to salbutamol after beta-blockers | 7-10 days
Incremental Shuttle Walk Test Result after taking beta-blockers | 7-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Bob Hancox, MD FRACP, Study Director — Waikato Hospital Research Unit
Locations (1):
- Department of Respiratory Medicine, Hamilton, Waikato Region, New Zealand